CLINICAL TRIAL: NCT01321411
Title: Clinical Respiratory Evaluation Using Spectroscopy Trial
Acronym: CREST
Status: Withdrawn | Type: Observational
Why Stopped: Not started and now discontinued
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-03356
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Respiratory Muscle Blood Flow
Keywords: Respiratory Muscle Blood Flow; Work of Breathing; Near Infrared Spectroscopy
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. ARDS/COPD: Critically ill patients with either ARDS or COPD weaning from mechanical ventilation.
  Interventions: Other: Near Infrared Spectroscopy
- 2. Healthy Volunteers
  Interventions: Other: Near Infrared Spectroscopy

INTERVENTIONS:
Other: Near Infrared Spectroscopy — Healthy Volunteers:
  Study #1 (Abnormal Pulmonary Resistance) subjects will breathe through a Starling resistor simulating abnormal pulmonary resistance. WOB and RMBF will be measured during resting breathing, as well as at 25%, 50% and 75% of MVV.
  Study #2 (Abnormal Pulmonary Compliance) subjects will breathe while wearing a chest binder simulating abnormal pulmonary resistance. WOB and RMBF will be measured during resting breathing, as well as at 25%, 50% and 75% of MVV.
  Groups: 2. Healthy Volunteers
Other: Near Infrared Spectroscopy — Clinical Volunteers:
  Study #3 (Abnormal Pulmonary Resistance) subjects recovering from COPD exacerbations will breathe through their ventilator circuit. PAV support will be altered to change the subjects' WOB. WOB and RMBF will be measured during resting breathing, as well as at 75%, 125% and 150% of baseline WOB.
  Study #4 (Abnormal Pulmonary Compliance) subjects recovering from ARDS will breathe through their ventilator circuit. PAV support will be altered to change the subjects' WOB. WOB and RMBF will be measured during resting breathing, as well as at 75%, 125% and 150% of baseline WOB.
  Groups: 1. ARDS/COPD

SUMMARY:
Respiratory muscles (the muscles used to breathe) need more blood (and oxygen) when their workload increases. It is difficult to measure respiratory muscle blood flow (RMBF) without invasive techniques. We will evaluate a new, much less invasive technique to measure RMBF in 2 groups: Healthy Volunteers and Critically Ill patients on breathing machines. The purpose of this study is to determine the accuracy of this new monitoring technique called Near Infrared Spectroscopy Utilizing Indocyanine Green Dye when compared with traditional measurements. The information gained from this study will help us to provide better care to patients with severe lung problems.

DETAILED DESCRIPTION:
PURPOSE To demonstrate the relationship between Respiratory Muscle Blood Flow and Work of Breathing using Near Infrared Spectroscopy utilizing Indocyanine Green Dye NIRS-ICG.

HYPOTHESIS AND OBJECTIVES

HYPOTHESIS #1: In subjects with normal respiratory muscle function (healthy volunteers) RMBF as measured by the NIRS-ICG technique will vary directly with work of breathing (WOB) as measured by changes in transpulmonary pressure gradients and as measured by Esophageal and Surface EMG.

Objective #1: To measure and demonstrate the relationship between RMBF and WOB/EMG in healthy volunteers simulating abnormal pulmonary resistance.

Objective #2: To measure and demonstrate the relationship between RMBF and WOB in healthy volunteers simulating abnormal pulmonary compliance.

HYPOTHESIS #2: In subjects with abnormal respiratory muscle function (weaning from mechanical ventilation after exacerbations of COPD or ARDS) RMBF as measured by the NIRS-ICG technique will vary with work of breathing as measured by changes in transpulmonary pressure gradients and as measured by Esophageal and Surface EMG.

Objective #3: To measure and demonstrate the relationship between RMBF and WOB in clinical subjects with abnormal pulmonary resistance (weaning from mechanical ventilation after COPD exacerbation).

Objective #4: To measure and demonstrate the relationship between RMBF and WOB in clinical subjects with abnormal pulmonary compliance (weaning from mechanical ventilation after ARDS).

HYPOTHESIS #3: We speculate, based on previous authors, that the blood flow rates in respiratory muscles for a given WOB will be different in clinical populations that in healthy volunteers. We hypothesize that the slope of the linear regression analysis relating BFI to WOB (both transpulmonary pressure gradients and EMG) will be "steeper" in clinical populations, suggesting that one reason for respiratory failure and weaning difficulties in these populations may be inefficient respiratory muscle oxygen utilization.

Objective #5: To demonstrate that the RMBF-WOB relationships in clinical populations will be different from that measured in healthy volunteers.

JUSTIFICATION To date, the measurement of regional blood flow and oxygen utilization has proven difficult. Nowhere is this more true than in the measurement of the regional blood flow and oxygen utilization of the respiratory muscles. Much of what we know about Respiratory Muscle Blood Flow (RMBF) stems from animal investigations or human research requiring highly invasive methods. The development of a minimally invasive technique for the measurement of RMBF has the potential to add significantly to our knowledge of respiratory energetics in research and clinical settings.

Near infrared spectroscopy (NIRS) can be used to measure the absorption of electromagnetic energy in the near infrared range (650 to 1000 nm) by in vivo chromophores. When assessing regional tissue oxygenation, NIRS assesses the amount of emitted energy absorbed in the range associated with hemoglobin (760 nm) and with deoxyhemoglobin (800 nm). The ratio of these amounts of absorbed light can be used to generate an index of tissue oxygenation/deoxygenation. Indocyanine green dye is a synthetic chromophore that absorbs energy in the infrared spectrum (805 nm). Guenette et al. measured the accumulation of ICG in respiratory muscles using NIRS while the concentration of ICG in the arterial blood was measured using photodensitometry. This technique has the advantage of being able to quantify absolute muscle blood flow with simultaneous measures of cardiac output, thereby allowing the calculation of absolute regional blood flows and absolute rates of regional oxygen uptake. The practicality of this technique in healthy volunteers is complicated by with the need for blood withdrawals and re-infusions as well as arterial cannulation and the measurement of cardiac output.

To avoid the logistical difficulties of arterial cannulation and central venous cannulation (required for the determination of cardiac output), a relative Blood Flow Index (BFI) has been proposed. The BFI method is a minimally invasive alternative and was first developed for rapid and repeated bedside estimation of cerebral blood flow. The BFI is derived from a transcutaneously measured NIRS ICG signal and does not require arterial cannulation or the measurement of cardiac output. BFI is a relative measure of blood flow as absolute flow cannot be determined unless arterial ICG concentration is measured.

Previous analyses have compared BFI and absolute muscle blood flow determined using NIRS and ICG and demonstrated strong agreement between BFI and NIRS derived absolute muscle blood flow. To date, no study has looked at the relationship between NIRS-ICG derived BFI values and respiratory workload as measured by esophageal and surface EMG (EEMG-SEMG) in subjects with abnormal compliance or resistance or in clinical populations.

Chronic Obstructive Pulmonary Disease (chronic bronchitis and emphysema), is a pathologic condition characterized by lung parenchyma destruction and abnormal airway narrowing that leads to a limitation of air. In clinical practice, COPD is defined by its characteristically low airflow and abnormal pulmonary system resistance during lung function tests. In contrast to asthma, this limitation is poorly reversible and progresses over time. COPD is the 4th leading cause of death amongst Canadians. Severe exacerbations of COPD may require mechanical ventilation and intensive care unit admission.

Acute Respiratory Distress Syndrome (ARDS) is a severe lung disease caused by both direct and indirect inflammatory injury. It is characterized by inflammation of the lung parenchyma leading to impaired gas exchange and abnormal respiratory system compliance. Hypoxemia and the release of systemically active cytokines frequently result in multiple organ failure and death. ARDS typically requires mechanical ventilation and admission to an intensive care unit.

Patients with COPD or ARDS that require mechanical ventilation are at high risk of death either from their disease or from complications during critical illness. Those that survive the acute phase of their illness often require prolonged mechanical ventilation and often have difficulty weaning from ventilator support. While lung parenchymal abnormalities and deconditioning are significant components of this "weaning failure", respiratory muscle strength, and potentially respiratory muscle blood flow, may play a role.

RESEARCH METHOD We will conduct a series of four studies to demonstrate the effectiveness of the Near Infrared Spectroscopy Indocyanine Green Dye (NIRS-ICG) technique for the non-invasive measurement of Respiratory Muscle Blood Flow (RMBF). The first two studies will occur in healthy volunteers and the second two studies will occur in clinical populations (mechanically ventilated patients recovering from exacerbations of COPD or recovering from ARDS). The first two studies will occur in our respiratory physiology laboratory (the Health and Integrative Physiology Laboratory at the University of British Columbia) and the second two will occur in the Intensive Care Unit (ICU) at VGH.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers

* 19 years of age or older
* Informed Consent Obtained
* No history of cardiopulmonary disease
* No history of smoking

Critically Ill

* 19 years of age or older
* Informed Consent Obtained
* Total pulmonary system resistance (as measured through the mechanical ventilator circuit) of 2-8 cmH20/L/second OR Total pulmonary system static compliance (as measured through the mechanical ventilator circuit) of 20-60 ml/cmH20

Exclusion Criteria for all studies:

* Esophageal lesions or esophageal surgery within the last 6 months
* Morbid obesity - defined as a Body Mass Index (BMI) > 40
* Allergy to any of the following: sulpha medications, penicillin, contrast dye, or iodine

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically Ill and Health Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Measure and demonstrate the relationship between RMBF and WOB | 3 hours
  To measure and demonstrate the relationship between RMBF and WOB in healthy volunteers simulating abnormal pulmonary resistance and compliance AND in critically ill subjects with abnormal respiratory muscle function (weaning from mechanical ventilation after exacerbations of COPD or ARDS).

SECONDARY OUTCOMES:
Demonstrate differences in RMBF-WOB between 2 cohorts | 3 hours
  We speculate that the blood flow rates in respiratory muscles for a given WOB will be different in clinical populations that in healthy volunteers.
  Objective: To demonstrate that the RMBF-WOB relationships in clinical populations will be different from that measured in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: William R Henderson, FRCPC, Principal Investigator — University of British Columbia